CLINICAL TRIAL: NCT07056218
Title: Outcome of RAI131 Therapy in Patients With Differentiated Thyroid Cancer (Low and Intermediate Risk)
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rana Ashraf Sabry, resident at oncology department nuclear medicine unit sohag university, Sohag University
Other Study IDs: Soh-Med-25-6-7MS
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low risk: patients typically have intrathyroidal papillary or follicular carcinoma, tumors <4 cm, no lymph node metastasis or only <5 small-volume (<0.2 cm) mico metastases, no vascular invasion (for follicular type), no aggressive histologic features, and no local or distant metastases.
  Interventions: Device: neck ultrasound; Diagnostic Test: thyroglobulin
- intermediate risk: includes cases with microscopic extrathyroidal extension (ETE), cervical lymph node metastases (especially >5 nodes or >0.2 cm), vascular invasion, aggressive histologic variants, or RAI-avid distant metastases
  Interventions: Device: neck ultrasound; Diagnostic Test: thyroglobulin

INTERVENTIONS:
Device: neck ultrasound — ultrasound scan
Diagnostic Test: thyroglobulin — blood test

SUMMARY:
Thyroid cancer is a universally relatively rare neoplasm, accounting for nearly 1-5% of all female cancers and less than 2% of male cancers. In spite of this relatively low incidence, it occupies the first rank among the most common endocrinal malignancies, with a consistent male to female ratio of 1: 3 observed in nearly all ethnic groups and geographic areas.

Differentiated thyroid cancer (DTC) is rated as slowly growing disease with a fairly good outcome where the five-year survival rate for localized tumor is 99.8% Total thyroidectomy, the removal of the entire thyroid gland, is the most common surgical approach-especially for tumors larger than 1 cm, multifocal disease, or suspected lymph node involvement. Lobectomy may be considered for small, low-risk tumors (<1 cm) confined to a single lobe. If lymph node metastasis is evident clinically or radiologically, neck dissection is performed. Postoperative radioactive iodine (RAI) therapy is used to ablate residual tissue or treat recurrent disease, particularly in iodine-avid tumors and intermediate- to high-risk patients. It may not be necessary for small, low-risk tumors. Thyroid hormone suppression therapy with levothyroxine serves both to replace thyroid hormone and suppress TSH, which could stimulate cancer growth. Long-term monitoring includes serial thyroglobulin (Tg) levels (along with anti-Tg antibodies if needed), neck ultrasound, and, in some cases, additional imaging like RAI scans or PET/CT to detect recurrence

ELIGIBILITY:
Inclusion Criteria:

- Pathologically or cytologically proven differentiated thyroid cancer.

* Total thyroidectomy with or without lymph node dissection
* Patient was treated by RAI after surgery
* Male and female patients
* Age >18 yrs

Exclusion Criteria:

* 1) Patients with undifferentiated thyroid cancer. 2) patients with high risk (distant metastasis) 3)patient with double malignancy 4) medullary thyroid cancer 4) Patient age < 18 years. 5)patient not treated by surgery or RAI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include 50 patients with thyroid cancer.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
outcome of radioactive iodine therapy on thyroid cancer | 12:18 months
  outcome of radioactive iodine therapy on thyroid cancer

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu Y, Su L, Xiao H. Review of Factors Related to the Thyroid Cancer Epidemic. Int J Endocrinol. 2017;2017:5308635. doi: 10.1155/2017/5308635. Epub 2017 May 2. PMID 28555155
- [Background] Baloch ZW, Asa SL, Barletta JA, Ghossein RA, Juhlin CC, Jung CK, LiVolsi VA, Papotti MG, Sobrinho-Simoes M, Tallini G, Mete O. Overview of the 2022 WHO Classification of Thyroid Neoplasms. Endocr Pathol. 2022 Mar;33(1):27-63. doi: 10.1007/s12022-022-09707-3. Epub 2022 Mar 14. PMID 35288841
- [Background] Tondi Resta I, Gubbiotti MA, Montone KT, Livolsi VA, Baloch ZW. Differentiated high grade thyroid carcinomas: Diagnostic consideration and clinical features. Hum Pathol. 2024 Feb;144:53-60. doi: 10.1016/j.humpath.2024.01.002. Epub 2024 Jan 19. PMID 38244615
- [Background] do Prado Padovani R, Duarte FB, Nascimento C. Current practice in intermediate risk differentiated thyroid cancer - a review. Rev Endocr Metab Disord. 2024 Feb;25(1):95-108. doi: 10.1007/s11154-023-09852-y. Epub 2023 Nov 23. PMID 37995023